CLINICAL TRIAL: NCT05522166
Title: The Effect of Digital Stories and Face-to-face Applied Basic Life Support Trainings on Knowledge and Skill Levels of Pre-service Teachers
Brief Title: Digital and Face-to-face Basic Life Support Training for Teacher Candidates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Uçar KÜÇÜK, Principal investigator, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KaradenizTechnical University
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Cardiopulmonary Resuscitation; Basic Life Support

STUDY DESIGN:
Intervention Model Description: The sample group determined by the stratified sampling method from the departments of the education faculty will be selected according to the simple random sampling method and distributed to the groups as 38 digital storytelling and 38 face-to-face applied training groups. In this pretest-posttest experimental study, data will be collected by using the student descriptive characteristics form, Basic Life Support Information Form and Basic Life Support Skills Evaluation Form in the pre-test. After the pre-test, BLS training will be carried out with digital storytelling for one group and face-to-face applied to the other group. The initiatives of both groups will last two months according to the program. After the training, post-test applications will be given to both groups. A permanence test will be given to both groups 1 month after the post-test.
Masking Description: Because the initiative of the study is based on the type of education. While obtaining informed consent, the purpose and content of the study were explained to the participants. For this reason, trainees know whether they will receive basic life support with digital storytelling or face-to-face applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Storytelling Group (Active Comparator): After the digital storytelling group teacher candidates are determined, forms and digital stories will be prepared to be used as pre-test, post-test and retention test. Afterwards, the skill assessment, in which the pre-test form will be applied, will be observed without intervention and evaluated by the researcher. Then, digital stories about TYD will be uploaded to social media for teacher candidates to watch. After watching these applications for two months, one-to-one applications will be made with teacher candidates in face-to-face education models. One month after the last test, the posttest and permanence test will be held in the same environment.
  Interventions: Other: Digital Stories and Face-to-face Basic Life Support Trainings
- Face to Face Applied Training Group (No Intervention): After the teacher candidates of the face-to-face application group are determined, the seminar training and program will be prepared. Then, the forms developed by the researcher will be applied as a pre-test. Pre-test skills of teacher candidates will be evaluated by the researcher with a skill evaluation form by making face-to-face observations on the model without any intervention. After the 8-week training of the teacher candidates is over, knowledge and skills will be given as a post-test. One month after the last test, retention tests will be done in a similar way.

INTERVENTIONS:
Other: Digital Stories and Face-to-face Basic Life Support Trainings — In this study, digital storytelling and face-to-face applied techniques will be given to teacher candidates via social media (Whatsapp) and the impact of these trainings on the knowledge and skill levels of teacher candidates will be evaluated comparatively.
  Arms: Digital Storytelling Group

SUMMARY:
Today, circulatory system and heart diseases, especially hypertension, are increasing day by day, and sudden and unexpected cardiac arrests due to these diseases are more common. Therefore, in the face of cardiac arrest that can develop without a certainty of time and place, Basic Life Support (TYD) is an important intervention that can save the lives of individuals with the least damage. Training on BLS, which is compulsory for healthcare professionals, is also given to some employees selected from other institutions. From this point of view, future teacher candidates who can be a role model in the society, at the same time reflect the importance of the subject to the group they work with and continue to teach, are an important group in terms of these trainings. Therefore, in this study, digital storytelling and face-to-face applied techniques will be given to teacher candidates via social media (Whatsapp) and the impact of these trainings on the knowledge and skill levels of teacher candidates will be evaluated comparatively.

DETAILED DESCRIPTION:
Purpose In order to develop knowledge and skills for a certain period of time, training is required for the BLS intervention to be performed in cases of cardiac arrest. It is important to provide BLS training for teachers who can reach a large part of the society. Therefore, it would be beneficial to train pre-service teachers on this subject during their education. BLS studies for teachers in the literature are generally limited to descriptive or one-time theoretical face-to-face trainings. This research is planned to evaluate the effects of digital stories and face-to-face applied basic life support training on the knowledge and skill levels of teacher candidates.

Method The universe of the research will consist of 711 pre-service teachers studying in the 3rd grade of Trabzon University teaching departments. The sample will consist of a total of 76 teacher candidates selected by power analysis. The sample group determined by the stratified sampling method from the departments of the education faculty will be selected according to the simple random sampling method and distributed to the groups as 38 digital storytelling and 38 face-to-face applied training groups. In this pretest-posttest experimental study, data will be collected by using the student descriptive characteristics form, Basic Life Support Information Form and Basic Life Support Skills Evaluation Form in the pre-test. After the pre-test, BLS training will be carried out with digital storytelling for one group and face-to-face applied to the other group. The initiatives of both groups will last two months according to the program. After the training, post-test applications will be given to both groups. A permanence test will be given to both groups 1 month after the post-test.

ELIGIBILITY:
Inclusion Criteria:

* Continuing education in the 3rd grade of the Faculty of Education of Trabzon University,
* To accept the work voluntarily,

Exclusion Criteria:

* Have a first aid instructor or trainer certification
* Studying at Trabzon University Faculty of Education 1st, 2nd and 4th Grades

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Student Identification Form | At the beginning of the study
  It was developed by the researcher based on the literature in order to define the socio-demographic characteristics of the pre-service teachers in both groups. The student introductory characteristics form consists of questions about the age, gender, marital status and reading part of the pre-service teachers.
Basic Life Support Information Form | up to 12 weeks
  The form will be developed by the researcher in order to determine the knowledge level of teacher candidates about basic life support based on the literature. This form, which will be used as a pre, post and retention test to measure the level of knowledge; anatomy of the respiratory and circulatory system, evaluation of vital signs, and basic life support. The forms will be filled by the teacher candidates. In the evaluation of the form, "yes" and "no" options will be used for correct answers and 1 point will be given for correct answers and 0 points will be given for wrong answers and I do not know.
Basic Life Support Skills Assessment Form | up to 12 weeks
  The form will be developed by the researcher in order to determine the skill level of teacher candidates regarding basic life support based on the literature. The form to be used as a pre, post and retention test to measure the skill level; It consists of questions with yes and no options questioning the process steps related to basic life support. The forms will be filled by observing the attempts made by the pre-service teachers after the skill attempts given. In the evaluation of the process steps, the pre-service teacher will be scored as "1" point for each correct step, and "0" point for each step that he/she does not/skip or erroneously/incompletely applies.
Preparation Phase of Digital Stories on Basic Life Support | up to 8 weeks
  In line with the Basic Life Support process steps, a total of 8 digital stories containing both knowledge and skills will be prepared. TYD information digital stories; 4 will be prepared on the anatomy of the respiratory and circulatory system, evaluation of vital signs, and basic life support. TYD Skill digital stories, on the other hand, will be prepared in 4 pieces, including the topics in the TYD skill form developed by the researcher.
Face to Face Applied Basic Life Support Seminar Training | up to 8 weeks
  This training; Ensuring scene safety, Evaluation of the situation, Detection of cardiac arrest, Activation of the emergency aid system, Performing effective and accurate heart compressions, Correct placement of the hands, Cardiac compression / rescue breath rate What to do for an effective compression, ensuring the opening of the airway and giving the rescue breath, Airway opening maneuvers will be prepared by the researcher based on the TYD guide on the Points to be Done on the training page of the Ministry of Health. Take into account the effective rescue breath, Recovery position.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want to share my individual participant data with other participants because I haven't completed my study yet.

REFERENCES:
- [Background] Mojtahedzadeh R, Mohammadi A, Hossein Emami A, Zarei A. How Digital Storytelling Applied in Health Profession Education: A Systematized Review. J Adv Med Educ Prof. 2021 Apr;9(2):63-78. doi: 10.30476/jamp.2021.87856.1326. PMID 34026906
- [Background] Rieger KL, West CH, Kenny A, Chooniedass R, Demczuk L, Mitchell KM, Chateau J, Scott SD. Digital storytelling as a method in health research: a systematic review protocol. Syst Rev. 2018 Mar 5;7(1):41. doi: 10.1186/s13643-018-0704-y. PMID 29506568
- [Background] Beck MS, Neil JA. Digital Storytelling: A Qualitative Study Exploring the Benefits, Challenges, and Solutions. Comput Inform Nurs. 2020 Jul 28;39(3):123-128. doi: 10.1097/CIN.0000000000000667. PMID 32732646
- [Background] Xie CY, Jia SL, He CZ. Training of Basic Life Support Among Lay Undergraduates: Development and Implementation of an Evidence-Based Protocol. Risk Manag Healthc Policy. 2020 Aug 5;13:1043-1053. doi: 10.2147/RMHP.S259956. eCollection 2020. PMID 32801977
- [Background] Martinez-Isasi S, Garcia-Suarez M, De La Pena Rodriguez MA, Gomez-Salgado J, Fernandez N, Mendez-Martinez C, Leon-Castelao E, Clemente-Vivancos A, Fernandez-Garcia D. Basic life support training programme in schools by school nurses: How long and how often to train? Medicine (Baltimore). 2021 Apr 2;100(13):e24819. doi: 10.1097/MD.0000000000024819. PMID 33787576
- [Background] Kim EJ, Roh YS. Competence-based training needs assessment for basic life support instructors. Nurs Health Sci. 2019 Jun;21(2):198-205. doi: 10.1111/nhs.12581. Epub 2018 Nov 15. PMID 30444071